CLINICAL TRIAL: NCT04325360
Title: Effects of Transcranial Direct Current Stimulation (tDCS) for the Treatment of Refractory Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Miriam Maria Pereira Novo, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18938319.7.0000.5404
Record Dates: First submitted 2019-12-10; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Epilepsy Intractable
Keywords: Epilepsy; transcranial direct current stimulation; seizures
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy; Seizures | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Prospective double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The tDCS machine is equipped with a sham option, determined by a code, that will not be disclosed to the participants, outcome assessor and principal investigator until the moment of data analysis. Randomization will be done through envelopes that will contain the codes of types of stimulation (real vs sham), which will be prepared by a third party.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cathodal Transcranial Direct Current Stimulation (c-tDCS) (Experimental): Participants in this arm of the study will receive cathode transcranial direct current stimulation.
  Interventions: Procedure: Cathodal Transcranial Direct Current Stimulation
- Sham-tDCS (Sham Comparator): Participants in this arm of the study will receive sham transcranial direct current stimulation.
  Interventions: Procedure: Sham Transcranial direct current stimulation

INTERVENTIONS:
Procedure: Cathodal Transcranial Direct Current Stimulation — 20 minutes of cathodal stimulation at 2mA, with cathode electrode placed over the focal epileptic area (determined by EEG exam and located according to the 10-20 system), the anode electrode will be placed over the supraorbital region, contralateral to the cathode electrode.
  Other Names: Transcranial direct current stimulation
  Arms: Cathodal Transcranial Direct Current Stimulation (c-tDCS)
Procedure: Sham Transcranial direct current stimulation — Participants will received 20 mins of Sham stimulation, where stimulation will happen for the first 30 seconds and in the last 30 seconds of the intervention (at 2mA), with no stimulation in the between time. The cathode electrode will be placed over the focal epileptic area (determined by EEG exam and located according to the 10-20 system),the anode electrode will be placed over the supraorbital region, contralateral to the cathode electrode.
  Arms: Sham-tDCS

SUMMARY:
The aim of this study is to investigate the effects of cathodal transcranial direct current stimulation in the management of seizures in subjects with focal refractory epilepsy.

DETAILED DESCRIPTION:
Hypothesis: Epilepsy is the most common neurological disorder globally, affecting approximately 50 million people worldwide. Of these, approximately 20% present with intractable or refractory epilepsy, where the frequency of seizures cannot be controlled adequately with anti-epileptic drugs (AEDs), leading to great neurobiological, cognitive, psychological and social consequences. Transcranial Direct Current Stimulation (tDCS) is a non-invasive brain stimulation (NIBS) technique that can effectively modulate (up- or down-regulate) cortical excitability of targeted brain regions. It has the potential of downregulating the neuronal activity, through the cathodal stimulation of the epileptic focal area and thus, reducing the frequency of seizures. Previous studies have shown that cathodal tDCS is a safe and effective treatment modality of treatment to reduce the frequency of seizures in patients with refractory epilepsy. However, the level of evidence of its effects in the management of seizures frequency is still low. In the present work, the investigators aim to evaluate the effects of tDCS in the management of seizures in patients with refractory epilepsy and its impact on cognitive function and quality of life.

Objective: The main aim of this randomized controlled trial is to determine if cathodal tDCS is effective in reducing the frequency of seizures in refractory epilepsy and, to determine if this reduction will positively impact the participants cognitive status and quality of life.

Methods: This is a prospective, randomized, placebo-controlled, double-blind, single-center study. The participants in the study will be randomized to either the intervention - tDCS group or sham group. Each individual will undergo 15 consecutive sessions of real cathodal tDCS stimulation or sham-stimulation. The primary outcome measure will be the frequency of seizures, measured by a seizure diary; changes in interictal epileptiform discharges on the Electroencephalogram (EEG); and functional connectivity changes in the epilepsy focal area, measured by resting-state Functional Resonance Image (rs-fMRI). Secondary outcomes include quality of life and cognition. Outcome measures will be done prior to intervention; immediately after intervention, at 1 month-follow up and again at 3-months follow up.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of focal refractory epilepsy
* participants must be 18 years or older
* must be on a stable medication regimen
* seizures frequency equal or greater than 1 seizure/month
* participants or their caregivers must be able to use a seizures diary

Exclusion Criteria:

* participants younger than 18 years old
* diagnosis of generalized epilepsy
* participants who are still making changes to medication regimen
* participants who are pregnant
* participants who have any kind of intracranial implants
* seizure frequency less than 1/month
* participants with skin abnormalities or rash on the scalp
* participants or caregivers that are unable to use a seizures diary

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in interictal epileptiform discharges on the electroencephalogram (EEG) | Pre-intervention, immediately post-intervention, 1 month post-intervention and 3 months post-intervention.
  EEG study will be conducted to determine changes in epileptiform discharge
Seizures Frequency | Pre-intervention, immediately post-intervention, 1 month post-intervention and 3 months post-intervention.
  Seizure frequency will be measured through the data analysis of a seizures diary
Changes in resting state connectivity through analysis of functional magnetic resonance imaging | Pre-intervention, post-intervention, 1 month post-intervention and 3 months post-intervention
  Resting state Functional Magnetic Resonance Image to determine changes in brain functional connectivity

SECONDARY OUTCOMES:
Changes in Cognitive function - Wechsler Adult Intelligence Scale (WAIS) | Pre-intervention, 1 month post-intervention, 3 months post-intervention
  Neuropsychological assessment to determine changes in attention, memory, executive functions skills
Positive changes in quality of life | Pre-intervention, 1 month post-intervention, 3 months post-intervention
  31-question questionnaire to determine quality of life changes specific to epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: Li Li Min, Study Director — University of Campinas, Brazil
Locations (1):
- Hospital das Clinicas - Unicamp, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No